CLINICAL TRIAL: NCT00490048
Title: Assessment of Pulmonary Involvement inUlcerative Colitis by Induced Sputum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hillel Yaffe Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ISUC.CTIL
Record Dates: First submitted 2007-06-21; First posted 2007-06-22 (Estimated); Last update posted 2007-06-22 (Estimated); Status verified 2007-06

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colits; lung; Induced sputum; Our aim to evaluate lung involvement in Ulcerative colitis patients by induced sputum
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Sodium Chloride

INTERVENTIONS:
Procedure: Induced sputum (inhalation of 3.5% saline)

SUMMARY:
Ulcerative colitis is a systemic disease we assume that extra intestinal involvement as we describein our study( Fireman Z, Osipov A, Kivity S, Kopelman Y, Sternberg A Fireman E: Assessment of pulmonary involvement in Crohn's disease by induced sputum. Am J Gastroenterol 2000;95(30):730-734. )

DETAILED DESCRIPTION:
Twenty Ulcerative colitis patients and 20 control subjects (all nonsmokers) without respiratory symptoms will be tested. The induce sputum by 20' inhalation of 3.5% saline using ultrasonic nebulizer. Samples will studied by differential counts of 200 cells on cytopreps stained by Giemsa. T-lymphocyte subset analyses were done by FACS using three monoclonal antibodies: CD3 = total T cells, CD4 = T helper cells, and CD8 = T suppressor-cytotoxic cells. CD4/CD8 >2.5 was considered abnormal.

ELIGIBILITY:
Inclusion Criteria:

* All the ulceratvive colitis patients without lung involvmentage 18-75 years of age

Exclusion Criteria:

* Pregnant women
* Non cooperative patients
* Smoker
* Lung disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
lung involvment in Ulcerative colitis patients

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Fireman, MD, Principal Investigator — Hillel- Yaffe Med. Ctr

REFERENCES:
- [Result] Fireman Z, Osipov A, Kivity S, Kopelman Y, Sternberg A, Lazarov E, Fireman E. The use of induced sputum in the assessment of pulmonary involvement in Crohn's disease. Am J Gastroenterol. 2000 Mar;95(3):730-4. doi: 10.1111/j.1572-0241.2000.01843.x. PMID 10710066